CLINICAL TRIAL: NCT01069601
Title: A Phase II Study to Evaluate the Immunogenicity, Safety and Tolerability of a H1N1 Influenza Vaccine in Immunocompromised Adults Who Have Undergone Solid Organ Transplantation or Bone Marrow Transplantation and in Age-Matched Healthy Volunteers
Brief Title: H1N1sw Vaccine in Adult Transplant Recipients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: End of H1N1 Swine Flu Pandemic
Sponsor: HepNet Study House, German Liverfoundation (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-017052-27; 200910H1N1MHH (Other: Hannover Medical School)
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Immunocompromised
Keywords: solid organ transplantation; bone marrow transplantation; adults; adults with solid organ transplantation; adults with bone marrow transplantation
MeSH Terms: interventions — focetria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- transplanted adults (Experimental): male and female adults who have previously undergone solid organ transplantation or allogeneic or autologous BMT
  Interventions: Biological: Focetria (2x H1N1 vaccine with MF59 adjuvants)

INTERVENTIONS:
Biological: Focetria (2x H1N1 vaccine with MF59 adjuvants) — 7,5µg H1N1sw monovalent vaccine with MF59 adjuvants; two doses 3 weeks apart
  Other Names: Focetria(R)

SUMMARY:
The trial investigates the efficacy of the adjuvanted H1N1 influenza vaccine Focetria(R) in immunocompromised adults who have undergone solid organ or bone marrow transplantation. It is expected that when administered twice the vaccine fulfills all serological efficacy criteria required for the elderly population age 60 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18-60 years of age who have undergone prior renal, cardiac, liver, lung, or bone marrow transplantation for any reason, more than 3 months prior to enrolment
* Patients able to visit the outpatient clinic with a life expectancy of at least one year
* Patients who receive any immunosuppressive treatment currently taken to prevent organ rejection

Exclusion Criteria:

* Individuals who received any vaccine within 30 days prior to study entry
* Individuals who received a H1N1 vaccination less than 6 months prior to the study
* Influenza diagnosed by a physician within 4 months prior to the study start
* Pregnant or lactating females
* History of an anaphylactic (i.e. life-threatening) reaction to any of the components of the vaccines, including egg and chicken proteins, ovalbumin, kanamycin and neomycin sulphate, formaldehyde and cetyltrimethylammonium bromide (CTAB)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The adjuvanted H1N1 influenza vaccine, when administered twice in transplanted patients, fulfils all serological efficacy criteria as required for the elderly population (aged 60 and older) according to the respective European guidance documents. | 42 days

SECONDARY OUTCOMES:
The adjuvanted H1N1 influenza vaccine in transplanted patients, when administered twice, is at least as effective as the adjuvanted H1N1 influenza vaccine in the healthy volunteers after only one administration. | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Manns, Prof, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany